CLINICAL TRIAL: NCT00494026
Title: Phase II Study of Concurrent Carboplatin, Pemetrexed, and Radiotherapy for Limited Stage of Small Cell Lung Cancer
Brief Title: Chemotherapy and Radiotherapy to Treat Patients With Limited Stage of Small Cell Lung Cancer (SCLC)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study stopped early based on interim results of another trial, showing inferior activity of pemetrexed/carboplatin compared to etoposide/carboplatin in SCLC.
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10015; H3E-MC-S095
Record Dates: First submitted 2007-06-27; First posted 2007-06-29 (Estimated); Results first posted 2009-11-17 (Estimated); Last update posted 2009-11-20 (Estimated); Status verified 2009-11

CONDITIONS: Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Pemetrexed; Carboplatin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pemetrexed + Carboplatin (Experimental)
  Interventions: Drug: pemetrexed; Drug: carboplatin; Procedure: radiotherapy

INTERVENTIONS:
Drug: pemetrexed — 500 milligrams per square meter (mg/m2), intravenous (IV), every 21 days x 2 cycles then 500 mg/m2, IV, every 21 days x 2 cycles
  Other Names: LY231514; Alimta
Drug: carboplatin — Area under the curve (AUC) 5, intravenous (IV), every 21 days x 2 cycles then AUC 5, IV, every 21 days x 2 cycles
Procedure: radiotherapy — 2 Gray (Gy) per fraction, 5 fractions per week, begin day 1, cycle 3 x 5 weeks (Monday-Friday)

SUMMARY:
This is a multicenter, phase II, open-label trial to evaluate the efficacy of pemetrexed + carboplatin combined with thoracic radiotherapy in patients with Limited Stage of small cell lung cancer

DETAILED DESCRIPTION:
Two 21-day cycles of pemetrexed (500 milligrams per square meter [mg/m2] intravenous [IV] infusion) and carboplatin (target area under the curve [AUC] 5 IV infusion) followed by two 21-day cycles of pemetrexed (500 mg/m2 IV infusion) and carboplatin (target AUC 5 IV infusion) with concurrent radiotherapy (2 Gray [Gy] per fraction, 5 fractions per week, up to a dose of 50 Gy is administered).

ELIGIBILITY:
Inclusion Criteria:

* Histologic and/or cytologic diagnosis of Limited Stage of small cell lung cancer
* Measurable disease
* Good performance status
* Adequate bone marrow reserve, hepatic, pulmonary and renal functions

Exclusion Criteria:

* Serious concomitant systemic disorder
* Prior chemotherapy for this cancer and/or prior thoracic radiotherapy
* Pregnancy/breast-feeding
* Significant weight loss over the previous 6 weeks before study entry
* Inability or unwillingness to take vitamin supplementation and corticosteroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2007-09; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (12):
- Italy (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orbassano
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Parma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Sisto
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Terni
- Poland (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Poznan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Warsaw
- Spain (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Palma de Mallorca
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Valencia
- United Kingdom (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Southampton, Hants
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guildford, Surrey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wolverhampton, West Midlands

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pemetrexed + Carboplatin
Started | 4
Completed | 0 (2 patients did receive the full study treatment prior to the study being terminated.)
Not Completed | 4
Not completed — Sponsor Decision | 4

BASELINE CHARACTERISTICS:
Arm/Group | Pemetrexed + Carboplatin
Number analyzed (Participants) | 4
Age Continuous [Mean (Standard Deviation); unit: years] | 59.85 (9.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 4
Region of Enrollment [Number; unit: participants]
  Poland | 2
  Spain | 2
Eastern Cooperative Oncology Group Performance Status [Number; unit: participants] — Classifies patients according to their functional impairment. Scores range from 0 (Fully Active) to 5 (Death).
  participants
    1 - Ambulatory, Restricted Strenuous Activity | 4
Race/Ethnicity [Number; unit: participants]
  Caucasian | 4

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With a Complete or Partial Response (Overall Response Rate [ORR])
Description: Overall Response Rate (ORR) was defined as the proportion of participants having either a Complete or Partial response using Response Evaluation Criteria In Solid Tumors (RECIST) criteria. Complete Response=disappearance of all target lesions; Partial Response=30% decrease in sum of longest diameter of target lesions.
Time Frame: baseline to measured response after chemotherapy and radiation
Population: Trial was stopped too early to assess the primary endpoint.
Measure: Number; unit: proportion of responders
Arm/Group | Pemetrexed + Carboplatin
Number analyzed (Participants) | 0

2. Secondary Outcome: Progression-free Survival
Description: Defined as the time from date of first dose to the first observation of disease progression, or death due to any cause.
Time Frame: baseline to measured progressive disease
Population: Trial was terminated early. Results were not analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed + Carboplatin
Number analyzed (Participants) | 0

3. Secondary Outcome: Overall Survival
Description: Overall survival is the duration from enrollment to death (includes 1 year follow-up). For patients who are alive, overall survival is censored at the last contact.
Time Frame: baseline to date of death from any cause, 1 year
Population: Trial was terminated early. Results were not analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed + Carboplatin
Number analyzed (Participants) | 0

4. Secondary Outcome: Duration of Response
Description: The duration of a complete response (CR) or partial response (PR) was defined as the time from first objective status assessment of CR or PR to the first time of progression or death as a result of any cause.
Time Frame: time of response to progressive disease
Population: Trial was terminated early. Results were not analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed + Carboplatin
Number analyzed (Participants) | 0

5. Secondary Outcome: Pharmacology Toxicity
Description: Radiation Therapy Oncology Group (RTOG) criteria were used for assessing toxicity. Toxicity grade reflected the most severe degree occurring during the evaluated period, not an average. When two criteria were available for similar toxicities, the one resulting in the more severe grade was used. Toxiccity grades range from 0 to 5. Toxicity grade = 5 if that toxicity caused the death of the patient.
Time Frame: every 21-day cycle for 4 cycles
Population: All enrolled patients who received radiotherapy.
Measure: Number; unit: participants
Arm/Group | Pemetrexed + Carboplatin
Number analyzed (Participants) | 2
participants
  Cycle 3: Grade 2 Hematologic White Blood Cell | 1
  Cycle 3: Grade 1 Platelets | 1
  Cycle 3: Grade 3 Neutrophils | 1
  Cycle 3: Grade 2 Hemoglobin | 1
  Cycle 3: Grade 2 Hematocrit | 1
  Cycle 4: Grade 3 Hematologic White Blood Cell | 1
  Cycle 4: Grade 3 Platelets | 1
  Cycle 4: Grade 2 Neutrophils | 1
  Cycle 4: Grade 3 Hemoglobin | 1
  Cycle 4: Grade 3 Hematocrit | 1

ADVERSE EVENTS:
Arm/Group | Pemetrexed + Carboplatin
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 2/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed + Carboplatin (N=4)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 2 (4)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (3)
Fatigue (General disorders) | 1 (1)
Mucosal inflammation (General disorders) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1)
Platelet count decreased (Investigations) | 2 (3)
Anorexia (Metabolism and nutrition disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days